CLINICAL TRIAL: NCT03410654
Title: Assessment of Cognitive Function Before and After Conversion From Immediate Release Tacrolimus to Envarsus XR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000022307; 000 (Other: CTGTY)
Record Dates: First submitted 2018-01-10; First posted 2018-01-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- adult kidney transplant recipients (Experimental): Adult kidney transplant recipients on tacrolimus immediate release for at least six months who are being converted to tacrolimus extended release Envarsus XR® (TAC XR) for any reason by a transplant nephrologist and are willing to participate in cognitive assessment will be offered the opportunity to participate in the study. An assessment is also made at the 3 month point as baseline.
  Interventions: Drug: Tacrolimus, Extended Release, (Envarsus Xr)

INTERVENTIONS:
Drug: Tacrolimus, Extended Release, (Envarsus Xr) — After conversion of tacrolimus immediate release to tacrolimus extended release.
  Other Names: Envarsus XR® (TAC XR)

SUMMARY:
The purpose of this study is to determine if cognitive function improves in patients converted from tacrolimus immediate release (TAC IR) to Envarsus XR® (tacrolimus extended release) using an objective measure of cognition.

DETAILED DESCRIPTION:
To assess cognitive function while on TAC IR and then three months after conversion to TAC XR using a traditional cognitive assessment, Montreal Cognitive Assessment (MoCA), and a broader cognitive assessment. This assessment will be used to determine if there is an objective improvement in cognitive function after conversion from TAC IR to TAC XR in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Post-renal transplant on stable TAC IR for at least 6 months who are converting to TAC XR regardless of indication.
* Patients receiving their post-transplant care through the Yale-New Haven Transplantation Center (YNHTC) regardless of where they were originally transplanted.

Exclusion Criteria:

* History of dementia or stroke
* Reside in a nursing home
* Newly started on an opiate, amphetamine, or benzodiazepine
* Non-English speaking (due to lack of NIH toolbox assessments in other languages)
* Patients that exhibit signs of acute infection, hemodynamic compromise or other signs of critical illness (e.g. respiratory distress requiring mechanical ventilation)
* Recipients of a multiorgan transplant
* Pregnant women
* Transplant recipients unable to provide informed consent to participate in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
cognitive assessment at baseline | baseline
  cognitive assessment at baseline using MoCA test 7.1
cognitive improvement from baseline | 3 months after enrollment
  cognitive evaluation from baseline average for adults using NIH Toolbox Cognitive Domain

SECONDARY OUTCOMES:
MoCA cognitive assessment | 3 months after enrollment
  cognitive assessment using MoCA 7.2
NIH Toolbox cognitive test | baseline
  NIH Toolbox Flanker Inhibitory Control and Attention Test
NIH Toolbox cognitive test | 3 months
  NIH Toolbox Flanker Inhibitory Control and Attention Test
NIH Toolbox cognitive test | baseline
  NIH Toolbox Dimensional Change Card Sort Test
NIH Toolbox cognitive test | 3 months
  NIH Toolbox Dimensional Change Card Sort Test
NIH Toolbox cognitive test | baseline
  NIH Toolbox Picture Sequence Memory Test Version A
NIH Toolbox cognitive test | 3 months
  NIH Toolbox Picture Sequence Memory Test Version B
NIH Toolbox cognitive test | baseline
  NIH Toolbox Pattern Comparison Processing Speed Test
NIH Toolbox cognitive test | 3 months
  NIH Toolbox Pattern Comparison Processing Speed Test
NIH Toolbox cognitive test | baseline
  NIH Toolbox List Sorting Working Memory Test
NIH Toolbox cognitive test | 3 months
  NIH Toolbox List Sorting Working Memory Test
NIH Toolbox cognitive test | baseline
  NIH Toolbox Reading Recognition Test
NIH Toolbox cognitive test | 3 months
  NIH Toolbox Reading Recognition Test

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cohen, PharmD, Principal Investigator — Yale New Haven Hospital; Richard Formica, MD, Principal Investigator — Yale Univeristy
Locations (1):
- Yale New Haven Transplantation Center, New Haven, Connecticut, United States